CLINICAL TRIAL: NCT06940388
Title: Total Neoadjuvant Treatment With or Without Tislelizumab for Locally Advanced Rectal Cancer: An Open-label Randomized Controlled Phase II Study (The TOTAL Trial)
Brief Title: Total Neoadjuvant Treatment With or Without Tislelizumab for Locally Advanced Rectal Cancer.
Acronym: TOTAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: brenner baruch (Other)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Sponsor-Investigator, brenner baruch, Head, Department of Oncology, Davidoff Cancer Center Rabin Medical Center, Beilinson Hospital Petach Tikva, Israel, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOTAL
Record Dates: First submitted 2025-04-01; First posted 2025-04-23 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Rectal Cancer (LARC)
Keywords: rectal cancer; locally advanced rectal cancer; total neoadjuvant treatment; immunotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-center, double arm, open-label, phase II randomized (1:1) controlled trial aimed to determine the efficacy and safety of TNT with or without tislelizumab in patients with primary, histologically proven LARC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TNT with Immunotherapy (Experimental): Patients will be treated with 6 weeks of capecitabine-based CRT followed 4 weeks later by 16 weeks of CIMT with tislelizumab and mFOLFOX6, both given Q2W.
  Interventions: Drug: Tislelizumab
- TNT (Other): Patients will be treated with 6 weeks of capecitabine-based CRT followed 4 weeks later by 16 weeks of chemotherapy with mFOLFOX6, Q2W.
  Interventions: Drug: Total neoadjuvant therapy (TNT)

INTERVENTIONS:
Drug: Tislelizumab — During ChemoImmunotherapy: Patients in the investigational arm will receive 8 cycles of tislelizumab 150 mg IV on Day 1, followed by mFOLFOX6 (Q2W).
  Arms: TNT with Immunotherapy
Drug: Total neoadjuvant therapy (TNT) — Patients will be treated with 6 weeks of capecitabine-based CRT followed 4 weeks later by 16 weeks of chemotherapy with mFOLFOX6, Q2W.
  Arms: TNT

SUMMARY:
This prospective, multi-center, phase II randomized controlled trial will evaluate the actual benefit of adding immunotherapy with tislelizumab to the currently most effective approach against LARC, namely TNT. In this trial, we will harness several elements that may each potentially contribute to an overall high efficacy, at least in local outcomes: nCRT rather than SCRT, full length (8 cycles of mFOLFOX6) of consolidation chemotherapy, CIMT following nCRT (exploiting the upregulation of the immune response induced by the latter) and tislelizumab (with its theoretical advantage over other CPIs). In line with the changing treatment paradigms in LARC, in which high therapeutic efficacy translates into the possibility to avoid TME, the trial will have a novel primary endpoint of long-term unmaintained cCR, i.e. 3 year TME-free survival.

DETAILED DESCRIPTION:
This is a prospective, multi-center, double arm, open-label, phase II randomized (1:1) controlled trial aimed to determine the efficacy and safety of TNT with or without tislelizumab in patients with primary, histologically proven LARC. All subjects will undergo a screening process, based on the inclusion and exclusion criteria listed below. All subjects confirmed to be eligible will be randomized (1:1) into one of the two study arms, using an eCRF software. Patients in the investigational arm will be treated with 6 weeks of capecitabine-based CRT followed 4 weeks later by 16 weeks of CIMT with tislelizumab and mFOLFOX6, both given Q2W. Patients in the control arm will be treated with 6 weeks of capecitabine-based CRT followed 4 weeks later by 16 weeks of chemotherapy with mFOLFOX6, without tislelizumab, Q2W. Patients in both arms will be re-staged 8 weeks (+/-14 days) after the completion of therapy. Patients who will achieve cCR/near cCR will be closely followed by WW, and will undergo TME at any sign of local tumor regrowth. Patients in both arms with residual tumor, will undergo immediate TME. All patients will be followed according to current NCCN guidelines.The primary aim of the trial is to demonstrate that an approach of adding tislelizumab to the chemotherapy phase of the neoadjuvant treatment will increase the 3 year TME-free survival rate by >20%, from 50% (based on the 53% 3 year TME-free survival rate in the OPRA trial) to 70% in patients with LARC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically confirmed primary (non-recurrent) LARC (tumor 12 cm or less from the anal verge, as assessed by rigid proctoscopy), stage T3-4 N0 or TX N+ according to base-line pelvic MRI and PET-CT.
* Patients who are planned for TNT and are surgical candidates as determined by the treating physician.
* No prior chemotherapy, immunotherapy, radiotherapy or surgery for rectal cancer.
* No prior radiotherapy to the pelvis, for any reason.
* Able to provide the FFPE block or 10 unstained slides from the colonoscopy for confirmation of the diagnosis, CPS status and for investigational purposes.
* Age 18 years or more.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) < 2.
* Screening laboratory values must meet the following criteria (using CTCAEv5.0):

  i) WBC > 2000/µL ii) Neutrophils > 1500/ µL iii) Platelets > 100 x 103/ µL iv) Hemoglobin > 9.0 g/dL v) Serum creatinine < 1.5 x ULN or calculated creatinine clearance > 60 mL/min (using the Cockcroft Gault formula) vi) AST and ALT < 2.5 x ULN. vii) Total bilirubin < 1.5 x ULN (total bilirubin must be < 3 x ULN for patients with Gilberts syndrome).
* Ability to swallow tablets.
* Adequate contraception in fertile patients; using a highly effective method of birth control for the duration of the study, and for at least 9 months after the last dose of chemotherapy and 120 days after the last dose of immunotherapy.
* Women of childbearing potential must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to the start of treatment.
* Women must not be breastfeeding.
* Signed written IRB approved informed consent. This must be obtained before the performance of any protocol related procedure that are not part of normal subject care. Subjects must be willing and able to comply with scheduled visits, treatments, and laboratory testing.

Exclusion Criteria:

* Active or background history of an autoimmune disease except for type I diabetes mellitus, hypothyroidism requiring hormone replacement only and skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment.
* Medical history of vasculitis.
* Prior organ transplant, including allogenic bone marrow transplantation.
* Grade > 1 peripheral sensory neuropathy.
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti- CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co- stimulation or checkpoint pathways.
* Any prior active malignancy < 2 years before trial entry except for any locally recurring cancer that has been treated curatively (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast).
* Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the subject to receive protocol therapy.
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Known acute hepatitis B, known chronic hepatitis B infection with active untreated disease, or known active hepatitis C infection. In participants with a history of HBV or HCV, participants with detectable viral loads will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
3-year total mesorectal excision (TME) free survival rates | Time from the date of registration to the date of TME or the first event of loco-regional failure, metastatic recurrence, the appearance of a secondary CRC or death from any cause. Assessed up to 36 months.
  3-year TME free survival will be defined as the percentage of patients who are alive and did not undergo total mesorectal excision (TME) surgery, or did not have an event of loco-regional failure, metastatic recurrence or the appearance of a secondary CRC, at 36 months of follow up.

SECONDARY OUTCOMES:
3 year TME-free survival rates of the CPS positive population | Time from the date of registration to the date of TME or the first event of loco-regional failure, metastatic recurrence, the appearance of a secondary CRC or death from any cause. Assessed up to 36 months.
  3-year TME free survival will be defined as the percentage of patients with CPS positive tumors (PDL-1 combined positive score >1%), who are alive and did not undergo total mesorectal excision (TME) surgery, or did not have an event of loco-regional failure, metastatic recurrence or the appearance of a secondary CRC, at 36 months of follow up.
Incidence of Treatment-Emergent Adverse Events (Safety) | Time from screening until the end of study drug administration, Immune-related AEs will be recorded up to 90 days (+7 days) after the last dose of tislelizumab. Assessed up to 11 months.
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0"
Disease-free survival (DFS) | Time from the date of registration to the date of the first event of loco-regional failure, metastatic recurrence, the appearance of a secondary CRC or death from any cause, assessed up to 36 months
  DFS will be censored for patients who are alive and free of progression at the time of last follow-up. DFS rate will be estimated using the Kaplan-Meier method
Overall survival (OS) | The time interval between the day of registration and the date of death of any cause, assessed up 60 months.
  Patients who are still alive when last traced will be censored at the date of last follow-up. OS rate will be estimated using the Kaplan-Meier method.
Progression-free survival (PFS) | The time from the date of registration to the date of the first objectively documented tumor progression, or death, whichever occurs first, assessed up to 60 months
  PFS is defined as the time from the date of registartion to the date of the first objectively documented tumor progression, or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (2):
- Johannes Gutenberg-University Clinic, Mainz, Germany 1.Dept. Medicine, Prof. Peter R. Galle, Mainz, Germany
- Davidoff Cancer Center, Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel RL, Miller KD, Fedewa SA, Ahnen DJ, Meester RGS, Barzi A, Jemal A. Colorectal cancer statistics, 2017. CA Cancer J Clin. 2017 May 6;67(3):177-193. doi: 10.3322/caac.21395. Epub 2017 Mar 1. PMID 28248415
- [Background] Siegel RL, Giaquinto AN, Jemal A. Cancer statistics, 2024. CA Cancer J Clin. 2024 Jan-Feb;74(1):12-49. doi: 10.3322/caac.21820. Epub 2024 Jan 17. PMID 38230766
- [Background] Bernier L, Balyasnikova S, Tait D, Brown G. Watch-and-Wait as a Therapeutic Strategy in Rectal Cancer. Curr Colorectal Cancer Rep. 2018;14(2):37-55. doi: 10.1007/s11888-018-0398-5. Epub 2018 Mar 7. PMID 29576755
- [Background] Zhong X, Wu Z, Gao P, Shi J, Sun J, Guo Z, Wang Z, Song Y. The efficacy of adding targeted agents to neoadjuvant therapy for locally advanced rectal cancer patients: a meta-analysis. Cancer Med. 2018 Mar;7(3):565-582. doi: 10.1002/cam4.1298. Epub 2018 Feb 21. PMID 29464874
- [Background] Habr-Gama A, Perez RO, Proscurshim I, Nunes Dos Santos RM, Kiss D, Gama-Rodrigues J, Cecconello I. Interval between surgery and neoadjuvant chemoradiation therapy for distal rectal cancer: does delayed surgery have an impact on outcome? Int J Radiat Oncol Biol Phys. 2008 Jul 15;71(4):1181-8. doi: 10.1016/j.ijrobp.2007.11.035. Epub 2008 Jan 30. PMID 18234443
- [Background] Garcia-Aguilar J, Chow OS, Smith DD, Marcet JE, Cataldo PA, Varma MG, Kumar AS, Oommen S, Coutsoftides T, Hunt SR, Stamos MJ, Ternent CA, Herzig DO, Fichera A, Polite BN, Dietz DW, Patil S, Avila K; Timing of Rectal Cancer Response to Chemoradiation Consortium. Effect of adding mFOLFOX6 after neoadjuvant chemoradiation in locally advanced rectal cancer: a multicentre, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):957-66. doi: 10.1016/S1470-2045(15)00004-2. Epub 2015 Jul 14. PMID 26187751
- [Background] Cercek A, Roxburgh CSD, Strombom P, Smith JJ, Temple LKF, Nash GM, Guillem JG, Paty PB, Yaeger R, Stadler ZK, Seier K, Gonen M, Segal NH, Reidy DL, Varghese A, Shia J, Vakiani E, Wu AJ, Crane CH, Gollub MJ, Garcia-Aguilar J, Saltz LB, Weiser MR. Adoption of Total Neoadjuvant Therapy for Locally Advanced Rectal Cancer. JAMA Oncol. 2018 Jun 14;4(6):e180071. doi: 10.1001/jamaoncol.2018.0071. Epub 2018 Jun 14. PMID 29566109
- [Background] Conroy T, Bosset JF, Etienne PL, Rio E, Francois E, Mesgouez-Nebout N, Vendrely V, Artignan X, Bouche O, Gargot D, Boige V, Bonichon-Lamichhane N, Louvet C, Morand C, de la Fouchardiere C, Lamfichekh N, Juzyna B, Jouffroy-Zeller C, Rullier E, Marchal F, Gourgou S, Castan F, Borg C; Unicancer Gastrointestinal Group and Partenariat de Recherche en Oncologie Digestive (PRODIGE) Group. Neoadjuvant chemotherapy with FOLFIRINOX and preoperative chemoradiotherapy for patients with locally advanced rectal cancer (UNICANCER-PRODIGE 23): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2021 May;22(5):702-715. doi: 10.1016/S1470-2045(21)00079-6. Epub 2021 Apr 13. PMID 33862000
- [Background] Galon J, Fridman WH, Pages F. The adaptive immunologic microenvironment in colorectal cancer: a novel perspective. Cancer Res. 2007 Mar 1;67(5):1883-6. doi: 10.1158/0008-5472.CAN-06-4806. PMID 17332313
- [Background] Nagtegaal ID, Marijnen CA, Kranenbarg EK, Mulder-Stapel A, Hermans J, van de Velde CJ, van Krieken JH. Local and distant recurrences in rectal cancer patients are predicted by the nonspecific immune response; specific immune response has only a systemic effect--a histopathological and immunohistochemical study. BMC Cancer. 2001;1:7. doi: 10.1186/1471-2407-1-7. Epub 2001 Jul 16. PMID 11481031
- [Background] Lin Z, Cai M, Zhang P, Li G, Liu T, Li X, Cai K, Nie X, Wang J, Liu J, Liu H, Zhang W, Gao J, Wu C, Wang L, Fan J, Zhang L, Wang Z, Hou Z, Ma C, Yang K, Wu G, Tao K, Zhang T. Phase II, single-arm trial of preoperative short-course radiotherapy followed by chemotherapy and camrelizumab in locally advanced rectal cancer. J Immunother Cancer. 2021 Nov;9(11):e003554. doi: 10.1136/jitc-2021-003554. PMID 34725214
- [Background] Zhang T, Song X, Xu L, Ma J, Zhang Y, Gong W, Zhang Y, Zhou X, Wang Z, Wang Y, Shi Y, Bai H, Liu N, Yang X, Cui X, Cao Y, Liu Q, Song J, Li Y, Tang Z, Guo M, Wang L, Li K. The binding of an anti-PD-1 antibody to FcgammaRIota has a profound impact on its biological functions. Cancer Immunol Immunother. 2018 Jul;67(7):1079-1090. doi: 10.1007/s00262-018-2160-x. Epub 2018 Apr 23. PMID 29687231
- [Background] Zitvogel L, Apetoh L, Ghiringhelli F, Kroemer G. Immunological aspects of cancer chemotherapy. Nat Rev Immunol. 2008 Jan;8(1):59-73. doi: 10.1038/nri2216. PMID 18097448
- [Background] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Lin ZY, Zhang P, Chi P, Xiao Y, Xu XM, Zhang AM, Qiu XF, Wu JX, Yuan Y, Wang ZN, Qu XJ, Li X, Nie X, Yang M, Cai KL, Zhang WK, Huang Y, Sun Z, Hou ZG, Ma C, Cheng FZ, Tao KX, Zhang T. Neoadjuvant short-course radiotherapy followed by camrelizumab and chemotherapy in locally advanced rectal cancer (UNION): early outcomes of a multicenter randomized phase III trial. Ann Oncol. 2024 Oct;35(10):882-891. doi: 10.1016/j.annonc.2024.06.015. Epub 2024 Jul 2. PMID 38964714
- [Background] Formenti SC, Demaria S. Systemic effects of local radiotherapy. Lancet Oncol. 2009 Jul;10(7):718-26. doi: 10.1016/S1470-2045(09)70082-8. PMID 19573801
- [Background] Goffredo P, Quezada-Diaz FF, Garcia-Aguilar J, Smith JJ. Non-Operative Management of Patients with Rectal Cancer: Lessons Learnt from the OPRA Trial. Cancers (Basel). 2022 Jun 30;14(13):3204. doi: 10.3390/cancers14133204. PMID 35804975